CLINICAL TRIAL: NCT00795704
Title: Effect of Mulberry Leaf Extract on Glycemic Durability in Non-insulin Dependent Diabetes Mellitus: a Double-blind, Randomized, Placebo-controlled Pilot Study (Mul-DM)
Brief Title: Impact of Mulberry Leaf on Type 2 Diabetes
Acronym: Mul-DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Riche, Assistant Professor of Pharmacy Practice and Medicine, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-0053
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: Herbal Supplement; Type 2 Diabetes; Mulberry; Hemoglobin A1C
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Morus alba

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Control Group
  Interventions: Drug: Placebo
- Mulberry Leaf Extract (Active Comparator)
  Interventions: Drug: Mulberry Leaf Extract

INTERVENTIONS:
Drug: Mulberry Leaf Extract — Mulberry Leaf Extract 1000 mg by mouth three times daily for 3 months
  Other Names: Mulberry; Morus indica L.; Morus alba
  Arms: Mulberry Leaf Extract
Drug: Placebo — Placebo 500 mg #2 capsules by mouth three times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether mulberry leaf extract will help control blood sugar in patients with type 2 diabetes. We also want to look at the safety of mulberry leaf extract in these patients.

DETAILED DESCRIPTION:
The methods for testing this hypothesis include: a 2-week placebo run-in, followed by a double-blind randomization into 2 groups: (1) mulberry leaf extract and (2) matching placebo. Evaluations of hemoglobin A1C (A1C) -- A measurement of blood glucose over the past 3 months -- will be done at baseline [before placebo run-in period] and 3 months. Evaluations of safety laboratories and adverse effect questionnaire will be done at 4 weeks and at 3 months following the randomization visit. Subjects will undergo a 2-week placebo run-in phase, and then will be divided into two groups: (1) mulberry leaf extract and (2) matching placebo. The subjects will ingest 1000 mg (#2 500 mg capsules) of standardized mulberry leaf extract (Nature-Gen, San Diego, CA) or matching placebo three times daily with meals for 3 months. Patients will be asked to monitor fasting morning blood glucose and 2-hour postprandial dinner blood glucose daily during the 2-week placebo run-in. To ensure compliance, only subjects compliant with both medication and monitoring instructions will be issued a 30-day supply of study medication at enrollment and the remainder at the 4-week safety visit. Each visit will consist of clinical examination, completed questionnaires, evaluation of self-monitoring blood glucose (SMBG), and donated blood for clinical laboratory tests. Standard recommendations for therapeutic lifestyle intervention will be given to both groups. All the clinical laboratory tests will be performed at the University of Mississippi Medical Center. All patients will receive identical 2-week placebo phase capsules, and then be randomized to each group using similar lookin

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* No diabetes medication adjustments for at least 2 months
* Stable hemoglobin A1C [Between 7.0% to 8.0% (inclusive) and not varying by more than 10% since prior visit; If no A1C exists prior to the current visit and no medication adjustments are made, the current A1C may used as the baseline]

Exclusion Criteria:

* On insulin
* History of overt cardiovascular disease
* History of missed appointments or non-compliance with medications
* History of hepatic or renal insufficiency
* History of hemoglobinopathies
* Women of reproductive potential not on oral contraceptives
* Pregnant/nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Riche, Pharm.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Andallu B, Varadacharyulu NC. Gluconeogenic substrates and hepatic gluconeogenic enzymes in streptozotocin-diabetic rats: effect of mulberry (Morus indica L.) leaves. J Med Food. 2007 Mar;10(1):41-8. doi: 10.1089/jmf.2005.034. PMID 17472465
- [Background] Mudra M, Ercan-Fang N, Zhong L, Furne J, Levitt M. Influence of mulberry leaf extract on the blood glucose and breath hydrogen response to ingestion of 75 g sucrose by type 2 diabetic and control subjects. Diabetes Care. 2007 May;30(5):1272-4. doi: 10.2337/dc06-2120. Epub 2007 Feb 15. No abstract available. PMID 17303787
- [Background] Hansawasdi C, Kawabata J. Alpha-glucosidase inhibitory effect of mulberry (Morus alba) leaves on Caco-2. Fitoterapia. 2006 Dec;77(7-8):568-73. doi: 10.1016/j.fitote.2006.09.003. Epub 2006 Sep 22. PMID 17071014
- [Background] Zhong L, Furne JK, Levitt MD. An extract of black, green, and mulberry teas causes malabsorption of carbohydrate but not of triacylglycerol in healthy volunteers. Am J Clin Nutr. 2006 Sep;84(3):551-5. doi: 10.1093/ajcn/84.3.551. PMID 16960168
- [Derived] Riche DM, Riche KD, East HE, Barrett EK, May WL. Impact of mulberry leaf extract on type 2 diabetes (Mul-DM): A randomized, placebo-controlled pilot study. Complement Ther Med. 2017 Jun;32:105-108. doi: 10.1016/j.ctim.2017.04.006. Epub 2017 Apr 27. PMID 28619294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruted from April 2008 - Feb 2010 in University of Mississippi Cardiometabolic clinic.
Pre-assignment Details: Two week placebo run-in
Groups:
- Mulberry Leaf Extract: 500 mg #2 capsules three times daily
Period: Overall Study
Arm/Group | Placebo | Mulberry Leaf Extract
Started | 12 | 12
Completed | 8 | 9
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mulberry Leaf Extract | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (7) | 57.3 (5.5) | 56.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Time Frame: 3 month minus baseline
Population: intention-to-treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | Mulberry Leaf Extract
Number analyzed (Participants) | 12 | 12
percent | -0.39 (0.51) | -0.26 (0.50)
Statistical Analysis 1: Comparison: Placebo vs Mulberry Leaf Extract; Test type: Superiority or Other; p = 0.079, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Adverse Drug Reactions, Abnormal Metabolic Panel Levels, or Abnormal Liver Enzyme Levels
Description: Sodium (>150 mmol/L), Potassium (>5 mmol/L), Bicarbonate (>34 mmol/L), Chloride (>110 mmol/L), Serum Creatinine (>1.2 mg/dL), Blood Urea Nitrogen (24 mg/dL), Calcium (>11 mg/L), Alanine Aminotransferase (>3 times baseline), Aspartate Aminotransferase (>3 times baseline) were collected at baseline, 1 month, and 3 months. Self-Reported adverse drug reactions are also reported.
Time Frame: Baseline, 1 month, and 3 months
Measure: Number; unit: participants
Arm/Group | Placebo | Mulberry Leaf Extract
Number analyzed (Participants) | 12 | 12
participants | 6 | 4

3. Secondary Outcome: Change From Baseline in Self-Monitoring Blood Glucose (SMBG) Averages
Description: 2-hour postprandial SMBG reported. A negative value indicates a decrease from baseline. A positive value indicates an increase from baseline.
Time Frame: Baseline and 3 months
Population: Intention-to-treat with data submitted baseline and final.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mulberry Leaf Extract
Number analyzed (Participants) | 6 | 8
mg/dL | -28.1 (36.3) | 3.6 (13.4)
Statistical Analysis 1: Comparison: Placebo vs Mulberry Leaf Extract; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 and 3 months
Arm/Group | Placebo | Mulberry Leaf Extract
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Mulberry Leaf Extract (N=12)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Warfarin intoxication after recent dose increase. Unrelated to study medication. Held study medication for 3 weeks per PCP, then resumed and completed.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Mulberry Leaf Extract (N=12)
GI Upset (Gastrointestinal disorders) | 3 (3) | 3 (4) — GERD, abdominal pain, gas, bloating, constipation
Allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — itching, watery eyes, sinus headache
Infection (Infections and infestations) | 2 (2) | 1 (1) — UTI, Influenza, skin infection
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No